CLINICAL TRIAL: NCT00971698
Title: The Spleen in Sickle Cell Anemia and Sickle Cell Thalassemia. Clinical Presentation and Follow up. Splenectomy, Indications and Complications.
Brief Title: The Spleen in Sickle Cell Anemia and Sickle Cell Thalassemia
Status: Completed | Type: Observational
Sponsor: HaEmek Medical Center, Israel (Other)
Responsible Party: Principal Investigator, Dr Koren Ariel, Head of Pediatric Hematology Unit and Pediatric Dpt B, HaEmek Medical Center, Israel
Other Study IDs: 0135-08-EMC
Record Dates: First submitted 2009-09-03; First posted 2009-09-04 (Estimated); Last update posted 2011-08-26 (Estimated); Status verified 2011-08

CONDITIONS: Sickle Cell Anemia; Thalassemia
Keywords: Splenectomy; Thrombocytosis; Infections; Spleen; Sickle Cell Thalassemia
MeSH Terms: conditions — Anemia, Sickle Cell; Thalassemia; Thrombocytosis; Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Sickle Cell Patients: Patients with homozygous Sickle Cell Anemia
- Sickle Cell Thalassemia: Patients with Sickle Cell Thalassemia

SUMMARY:
The spleen in Sickle Cell Anemia and Sickle Cell Thalassemia is usually enlarged in the first years of life but the immune protection provided is considered insufficient. In homozygous Sickle cell patients the spleen usually developed recurrent infarcts and after the first decade of age become fibrotic. Acute splenic sequestration is also frequent in those patients and this is considered as an indication for splenectomy.

In comparison in Sickle cell thalassemia patients, hypersplenism is more frequent.

The purpose of this study is to compare the clinical and laboratory issues related to the spleen in two groups of Sickle cell patients.

DETAILED DESCRIPTION:
Clinical and laboratory characteristics related to the spleen in SCA patients will be studied.

Two groups of patient will be compared, a group of Sickle cell patients (Homozygous) and a second group of patients with Sickle cell beta thalassemia.

In those patients that splenectomy was performed the incidence of infections will be recorded besides the indications for splenectomy and the incidence of thrombotic events or thrombocytosis.

ELIGIBILITY:
Inclusion Criteria:

* All the patients followed up at the Pediatric Hematology Unit

Exclusion Criteria:

* Patients lost from follow up of with insufficient data

Ages: 1 Year to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Two groups of patients: 25 patients with homozygous Sickle Cell Anemia and 25 patients with Sickle Cell Thalassemia
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2009-02; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Clinical events and abnormal laboratory results | One year

CONTACTS AND LOCATIONS:
Locations (1):
- Pediatric Hematology Unit and Pediatric Dpt B - HaEmek Medical Center, Afula, Israel